CLINICAL TRIAL: NCT05430607
Title: The Impact of Running Therapy on Mental Health of Youth in the In-patient and Daycare Centers of the Psychiatric Adolescent Department, Ziv Medical Center, Safed - A Pilot Randomized Controlled Trial
Brief Title: The Impact of Running Therapy on Mental Health of Youth in a Psychiatric Adolescent Department
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tali Bertler (Other Government)
Responsible Party: Sponsor-Investigator, Tali Bertler, Principal Investigator, Ziv Hospital
Organization: Ziv Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0119-21-ZIV
Record Dates: First submitted 2022-04-05; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Psychiatric Disorder; Mental Health Issue
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: 2 parallel study arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will participate in a 9-week running program and will also continue their routine treatment program at the psychiatric ward.
  Interventions: Behavioral: Running therapy
- Control group (No Intervention): The control group will continue their routine treatment program at the psychiatric ward.

INTERVENTIONS:
Behavioral: Running therapy — A 9-week running program.
  Arms: Intervention group

SUMMARY:
A randomized controlled trial, whereby the intervention group will participate in a 12-week running program and will also continue their routine treatment program. The control group will continue the treatment program as usual.

DETAILED DESCRIPTION:
Patients in the inpatient and daycare centers of the psychiatric adolescent department at Ziv Medical Center receive an intensive treatment program including medical management, psychotherapy (individual, groups, and family therapy), and suited educational and other extracurricular recreational activities. Despite growing evidence of the effective influence of aerobic physical activity and running therapy, it is not included in the intensive treatment program, and, as far as we know, it is not included in most psychiatric wards in Israel.

The aim of this study is to assess the effectiveness of combining a group based running therapy as part of the treatment program provided in the inpatient and day care centers of the psychiatric ward.

A randomized controlled trial, whereby the intervention group will participate in a 12-week running program and will also continue their routine treatment program. The control group will continue the treatment program as usual.

Participants will have group running sessions for 1 hour, three times a week, for 12 weeks. Sessions will include a psycho-educational short explanation, warm-up, main running exercise, relaxation, and a short summing up discussion. The sessions will be at an open court near the hospital. It will be guided by a team that will address both physical and therapeutic aspects.

The intervention program will include running outside the hospital complex (Safed Stadium) 3 times a week for about an hour each time, for 12 weeks. Participants will be transported to the stadium in an organized manner where the therapeutic running training will be conducted by a team that will include the researcher, running coach, nursing staff and psychology students.

Sessions will include a psycho-educational short explanation, warm-up, main running exercise, relaxation, and a short summing up discussion. At the end of the session, the participants will be driven back to the inpatient ward and day care centers.

Participants from the intervention group will be given specific group running T-shirts. Every week they will be given motivation band bracelets. The control group will be given similar items. Also, both groups will be given running shoes.

ELIGIBILITY:
Inclusion Criteria:

* 12-18-year-olds.
* Expected to be under observation for at least 10 weeks at time of recruitment.
* Consent of the patients and their parents to participate in the randomized control trial

Exclusion Criteria:

* Acute psychosis or manic states
* Acute suicidality
* Extreme physical difficulties
* Anorexia Nervosa

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms | 1-2 weeks before the start of the intervention and at the end of the intervention (10-11 weeks after the start of the intervention)
  Depressive status will be measured using the Children Depression Inventory (CDI; Kovacs, 1992) before and after the intervention to assess the change in symptoms.
Change in anxiety symptoms | 1-2 weeks before the start of the intervention and at the end of the intervention (10-11 weeks after the start of the intervention)
  Anxiety level will be measured by Screen for Child Anxiety Related Emotional Disorders (SCARED; Birmaher et al., 1997, 1999) before and after the intervention to assess the change in symptoms.

SECONDARY OUTCOMES:
Change in self compassion symptoms | 1-2 weeks before the start of the intervention and at the end of the intervention (10-11 weeks after the start of the intervention)
  Self-compassion will be measured by The Self-Compassion Scale-Short Form (SCS-SF; Raes, Pommier, Neff, & Van Gucht, 2011) before and after the intervention to assess the change in symptoms.
Change in emotion regulation symptoms | 1-2 weeks before the start of the intervention and at the end of the intervention (10-11 weeks after the start of the intervention)
  Emotion dysregulation will be measured by16-item version of the Difficulty in Emotion Regulation Scale (DERS-16; Bjureberg et al., 2016) before and after the intervention to assess the change in symptoms.
Change in self-efficacy symptoms | 1-2 weeks before the start of the intervention and at the end of the intervention (10-11 weeks after the start of the intervention)
  Self-Efficacy will be measured by the 10 item General Self Efficacy Scale (GSES; Schwarzer, & Jerusalem, 1979, 1981, 1995) before and after the intervention to assess the change in symptoms.
self injurious behavior | 1-2 weeks before the start of the intervention and at the end of the intervention (10-11 weeks after the start of the intervention)
  Self-injury will be measured by Direct self-injurious behaviors (D-SIB, i.e., selfinjury) before and after the intervention to assess the change in symptoms.

OTHER OUTCOMES:
therapeutic components' effect on mental health | 10-11 weeks after the start of the intervention (at the end of intervention).
  A specially designed questionnaire will address the effect on the therapeutic relationship and satisfaction that will include aspects of therapeutic alliance with the therapist, group aspects of treatment and the physical parts from the run itself.

CONTACTS AND LOCATIONS:
Overall Officials: Tali Bertler, PhD, Principal Investigator — Ziv Medical Center
Locations (1):
- Psychiatric adolescent department, Ziv Medical Center, Safed, Israel

IPD SHARING:
Plan to Share IPD: No